CLINICAL TRIAL: NCT05574244
Title: Comparison of Functional Outcomes of Ejaculation-preserving Partial Trans Urethral Resection of the Prostate With Complete Trans Urethral Resection of the Prostate for Benign Prostatic Obstruction
Acronym: PARTURP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: CHUBX 2019/57
Record Dates: First submitted 2022-09-13; First posted 2022-10-10 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-06

CONDITIONS: Benign Prostatic Hyperplasia
Keywords: Lower Urinary Tract Symptoms; Transurethral resection of prostate; Partial Transurethral resection of prostate; quality of life; Ejaculation
MeSH Terms: conditions — Prostatic Hyperplasia; Lower Urinary Tract Symptoms

STUDY DESIGN:
Intervention Model Description: Non inferiority Comparative single-blinded (patient) multicentre randomised clinical trial in two parallel groups:
  * Group 1: Conventional endoscopic prostatic surgery
  * Group 2: Partial surgery preserving the prostatic apex
Who Masked: Participant
Masking Description: * The clinical research assistant will fill-out the electronic case report form (eCRF) "randomisation" page and perform the randomisation. The site will immediately provide the study identification number for the patient and the allocation group.
  * The clinical research assistant will print the result of the randomisation. The printed document will be placed in a sealed envelope that will be stored in the patient's file.
  * The surgeon will open the envelope in the operating theatre once the patient has been placed under general anaesthesia.
  To prevent breaking the blinding post-operatively, the complete or partial aspect of endoscopic resection will not be mentioned in the surgical report (the patient will be specifically informed of that particular point before signing the informed consent). The complete or partial aspect of surgery will be revealed to patients at the end of follow-up, and in case of any surgical problem (e.g. need for re-intervention) or consent withdrawal.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional endoscopic prostatic surgery (Experimental): Endoscopic resection of prostate.
  Interventions: Procedure: Conventional endoscopic prostatic surgery
- Partial surgery preserving the prostatic apex (Experimental): Patients randomised to the partial endoscopic resection group will undergo surgical treatment that preserves the apex area of the prostate (tissue located 1 cm around the veru montanum).
  Interventions: Procedure: Partial surgery preserving the prostatic apex

INTERVENTIONS:
Procedure: Partial surgery preserving the prostatic apex — Partial Endoscopic resection of prostate to conserve apex
  Arms: Partial surgery preserving the prostatic apex
Procedure: Conventional endoscopic prostatic surgery — Endoscopic resection of prostate.
  Arms: Conventional endoscopic prostatic surgery

SUMMARY:
It has been demonstrated that sexual activity was common in the majority of men over 50 years old and was an important component of overall quality of life (QoL). Ejaculatory dysfunction (EjD) is the most common side effect of surgical treatment of benign prostatic obstruction (BPO). It has been considered for decades to be an inevitable consequence of restoring micturition comfort. EjD can have a substantial deleterious effect on the QoL of men with previously maintained regular sexual activity, inducing decreased orgasmic intensity and increased levels of anxiety and depression. A better understanding of the physiology of ejaculation has enabled the emergence of modified surgical techniques that aim to preserve antegrade ejaculation. Our hypothesis is that conservation of ejaculation can be achieved by modified surgical procedures without compromising functional outcomes.

DETAILED DESCRIPTION:
The aim of this study is To compare the efficacy of partial trans urethral resection of the prostate versus conventional resection of the prostate in improvement of lower urinary tract symptoms related to benign prostatic hyperplasia at 6 months. The secondary objectives are to compare the impacts of partial prostatic endoscopic surgery versus conventional endoscopic surgery on ejaculatory function, lower urinary tract symptoms, Global sexual life, Urinary flow, complication related to the surgery and the rates of re-treatment.

Investigators use a non-inferiority comparative single blinded (patient) multicenter randomized clinical trial in two parallel groups (Conventional endoscopic prostatic surgery Vs Partial surgery preserving the prostatic apex.

ELIGIBILITY:
Inclusion Criteria:

* Man over 40 years old
* Indication of surgical management for BPH
* Prostate volume ≥30 cc and ≤150 cc as evaluated by ultrasonography ( or an MRI if available)
* IPSS score ≥12
* Qmax ≤15 ml/s
* Affiliated to French national social security system
* wish and be able to comply with planned visits
* Able to express his consent
* Signed informed consent form

Exclusion Criteria:

* Unwillingness to accept the treatment
* No pre-operative ejaculation or sexuality
* Neurological pathology responsible for micturition disorders
* History of prostatic surgery
* Stenosis of the urethra symptomatic
* History of prostate cancer
* History of radiotherapy or pelvic surgery
* Patient refusing the principle of partial surgery
* Life expectancy <3 years
* Inability to understand the informed consent document, to give consent voluntarily or to complete the study tasks.
* Participation in another clinical study involving an investigational product within 1 month before study entry.

Min Age: 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Man over 40 years old
Enrollment: 336 (Estimated)
Dates: Start 2022-09-29 (Actual); Primary Completion 2029-03-31 (Estimated); Study Completion 2029-03-31 (Estimated)

PRIMARY OUTCOMES:
Evaluation of IPSS (International Prostatic Symptom Score) score at 6 months | 6 months after surgery
  the mean IPSS score measured at 6 months, to compare the efficacy of partial endoscopic resection versus complete endoscopic resection in improvement of lower urinary tract symptoms related to BPH. IPSS scores are categorised as 'asymptomatic' (0 points), 'mildly symptomatic' (1-7 points), 'moderately symptomatic' (8-19 points), and 'severely symptomatic' (20-35 points).

SECONDARY OUTCOMES:
Evaluation of ejaculation and global sexual life | 1 month, 3 months, 6 months,12 months, and 36 months after surgery
  MSHQ ejd= Male Sexual Health Questionnaire for Ejaculatory Dysfonction Scale score : [1-20] : a higher score mean that the subject have a ejaculatory dysfunction and sexual troubles
Evaluation of lower urinary tract symptoms | 1 month, 3 months, 6 months,12 months, and 36 months after surgery
  Urinary Symptom Profile (USP) :
  * 1a+1b+1C [0-9]. A higher score mean that the subject have urinary leakage
  * 2+3+4+4bis+5+6+7 [0-21]. A higher score mean that the subject have voiding urgency
  * 8+9+10 [0-9]. A higher score mean that the subject have voiding problem
Evaluation of complication rates | 1 month, 3 months, 6 months,12 months, and 36 months after surgery
  Complications based on Clavien Dindo classification
Evaluation of ejaculation and global sexual life | 1 month, 3 months, 6 months,12 months, and 36 months after surgery
  IIEF-15 (including orgasmic function: questions 9 and 10), auto-questionnaire (superiority test)
Evaluation of ejaculation and global sexual life | 1 month, 3 months, 6 months,12 months, and 36 months after surgery
  DAN PPS-SEX= Danish Prostatic Symptom Score -Sexual Questions 1A And B are question about erectyl function Questions 2A, 2B, 3A and 3B are questions about ejaculatory function Questions 4A is a question about global sexual quality of life
Evaluation of lower urinary tract symptoms | 1 month, 3 months, 6 months,12 months, and 36 months after surgery
  IPSS = International Prostate Score Symptom Scale score [0-35]. The higher score mean that the subject have important lower urinary tract symptoms.
Evaluation of lower urinary tract symptoms | 1 month, 3 months, 6 months,12 months, and 36 months after surgery
  Qmax (non-inferiority test) not performed at 1 month
Evaluation of complication rates | 1 month, 3 months, 6 months,12 months, and 36 months after surgery
  Re-intervention rate

CONTACTS AND LOCATIONS:
Locations (18):
- France (18):
  - CH Pays d'Aix, Aix-en-Provence
  - CHU Angers, Angers
  - Centre Hospitalier Universitaire de Bordeaux, Bordeaux
  - CHU Mondor, Créteil
  - Hôpital Claude Huriez, Lille
  - CHU de Limoges, Limoges
  - Hôpital Nord Marseille, Marseille
  - Polyclinique Saint George, Nice
  - Hôpital cochin, Paris
  - Hôpital Prive Francheville, Périgueux
  - Hôpital Lyon Sud HCl Bât.3C Centre Hospitalier Lyon Sud, Pierre-Bénite
  - Hôpital Privé des Côtes D'Armor, Plérin
  - CHU de Reims- Hôpital Robert Debré, Rennes
  - CHU de Rennes Pontchaillou, Rennes
  - CHU de Rennes, Rennes
  - Clinique Pasteur, Toulouse
  - CHRU Hôpitaux de tours, Tours
  - Hopital Privé de Versailles, Clinique des Franciscaines, Versailles

IPD SHARING:
Plan to Share IPD: No